CLINICAL TRIAL: NCT04873674
Title: A Deep Learning Algorithm Platform to Predict Autism Diagnosis and Subtypes by Integrating Clinical, Cognitive, Imaging, Gut Microbiome, and Metabolome Data
Brief Title: A Deep Learning Algorithm Platform to Predict Autism Diagnosis and Subtypes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002086RIND
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — metabolite (blood) and intestinal microbial (stool)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASD group: 240 ASD patients (aged 4-25 years)
  Interventions: Other: ASD diagnosis; Other: Psychiatric diagnosis
- Unaffected siblings of ASD: 60-100 unaffected siblings of ASD probands
  Interventions: Other: Psychiatric diagnosis
- TD group: 120 age-, and sex matched TDC from the same geographic areas of the ASD group via referral by teachers, or advertisement at college or community.
  Interventions: Other: Psychiatric diagnosis

INTERVENTIONS:
Other: ASD diagnosis — Autism Diagnostic Interview-revised (ADI-R) and Autism Diagnostic Observation Scale (ADOS)
  Groups: ASD group
Other: Psychiatric diagnosis — Kiddie Schedule for Affective Disorders & Schizophrenia (K-SADS) for DSM-5

SUMMARY:
This is the first human study on ASD microbiome with robust methodologies: prospective and sibling designs, metagenomics profiles, establishing an ASD multi-dimensional databank (clinic, behavior, neurocognition, brain imaging, metabolomics, and microbiome) collected using the same methodology and genetic biology simultaneously, and developing a deep learning platform for ASD diagnosis and prevention. With the accomplishment of this project, we anticipate establishing a web application for clinical and academic use. Our findings will further advance the knowledge in the pathogenetic mechanisms of ASD to enhance early detection, diagnosis, and treatment, subsequently contributing to precision medicine.

DETAILED DESCRIPTION:
Due to the high prevalence (1% in Taiwan), long-lasting impairment, unclear etiologies, and a lack of effective detection, prevention, and biological treatment, autism spectrum disorder (ASD) has been prioritized for biomarker, mechanism, and treatment research. Recently the gut-brain-axis has been proved, mainly with animal models, to be altered in psychiatric disorders and notably in ASD. With PI Gau's long-term achievement in ASD multi-dimensional research and our preliminary finding of altered gut microbiota in ASD and their unaffected siblings, we propose this 4-year prospective large-scale study with sibling design and multi-dimensional measures (environmental, clinical, cognitive, imaging, gut microbiome, metabolome) to establish a deep learning algorithm platform for predicting ASD and searching potential biomarkers and probiotic treatment for ASD.

Specific Aims:

1. To demonstrate the metagenomics profiles analysis based on the gut microbiome and metabolome of ASD patients, unaffected siblings, and typically developing controls (TDC).
2. To investigate environmental factors such as pregnancy and birth history from the mother's medical records and interviews or national health insurance data, for the microbiome, metagenomics, and brain anatomy and function.
3. To develop a deep learning algorithm platform using the environmental, behavioral/clinical phenotypes, neurocognitive/imaging endophenotypes, and metagenomics profiles to identify microbiota (metagenomics, too) makers and other predictors for ASD diagnosis, subtypes, and level of impairments.
4. To establish a web application based on our deep learning algorithm platform for clinical use to assist medical doctors in diagnosing ASD.

ELIGIBILITY:
Inclusion Criteria:

* ASD participants are (1) they have a clinical diagnosis of ASD defined by the DSM-5 criteria,1 made by board-certificated child psychiatrists and confirmed by the ADI-R/ADOS; (2) their ages range from 4 to 25; (3) both parents are Han Chinese; (4) they and their parents cooperate with all the assessments and stool and blood collection.

Inclusion Criteria for US and TDC are (1) they do not reach the clinical diagnosis of ASD according to DSM-5 diagnostic criteria and the same criteria as described in the (2), (3), (4) and of Inclusion Criteria for ASD participants.

Exclusion Criteria:

* (1) comorbidity with DSM-5 diagnoses of schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorders, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use; (2) comorbidity with neurological or systemic disorders; and (3) having a first degree relative who may have ASD based on family history method assessment (the TDC group).

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample includes 240 ASD (aged 4 to 25 years), 60~100 (estimated average 80) unaffected siblings (US), and 120 TDC. 240 ASD and 80 US, aged 4-25 will be recruited from the ASD follow-up cohort established by PI Gau's NHRI project or the Department of Psychiatry of all the branches of NTUH.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Autism diagnostic interview (ADI-R) | 4 hours
  Including reciprocal social interaction, communication, and repetitive behaviors and stereotyped patterns, for children with a mental age from about 18 months into adulthood
Neuropsychological functions: Continuous Performance Test(CPT) | 15 minutes
  The 4 dimensions of CCPT: focused attention, hyperactivity/impulsivity, sustained attention, and vigilance
Neuropsychological functions: Cambridge Neuropsychological Test Automated Batteries(CANTAB) | 1.5 hours
  The 4 main cognitive components of CANTAB: Visual Memory, Attention, Working and Planning Memory (Executive Functions), and Decision Making

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan